CLINICAL TRIAL: NCT01977807
Title: A Prospective Safety and Effectiveness Study of the 500 Hz Technolas Perfect Vision Excimer Laser in Asian Eyes Using LASIK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1303
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Myopia; Hyperopia; Presbyopia
Keywords: Myopia; Hyperopia; Presbyopia; Supracor; Zyoptix; Proscan; LASIK
MeSH Terms: conditions — Myopia; Hyperopia; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Myopia (Experimental): Myopia Lasik treatment of virgin eyes.
  Interventions: Device: Proscan, Zyoptix and Supracor
- Hyperopia (Experimental): Hyperopia Lasik treatment of virgin eyes.
  Interventions: Device: Proscan, Zyoptix and Supracor

INTERVENTIONS:
Device: Proscan, Zyoptix and Supracor — One device (500 Hz Excimer Laser) with three interventions (Proscan, Zyoptix and Supracor as algorithms)

SUMMARY:
This clinical study has been planned to evaluate the safety and effectiveness of common treatment algorithms using 500 Hz laser repetition rate.

DETAILED DESCRIPTION:
This clinical study has been planned to evaluate the safety and effectiveness of the excimer laser treatment algorithms Proscan, Zyoptix and Supracor of the 500 Hz laser system for ametropia and/or presbyopia when performed on the cornea of virgin eyes.

ELIGIBILITY:
General Inclusion Criteria

* Subjects have to be at least 18 years of age.
* Subjects have to be able to read, understand, and sign a statement of Informed Consent.
* Subjects have to be willing and able to return for scheduled follow-up examinations for up to 6 and 12 months respectively after surgery.
* Corneal topography should be qualified
* High contrast, manifest, best spectacle-corrected distance visual acuity correctable binocular to at least 1.0 (Snellen 20/20 or 6/6) and monocular to at least 0.8 (Snellen 20/25 or 6/7.5). In case of a monocular surgery the eye which should not be treated must have a best corrected distance visual acuity of at least 0.8 (Snellen 20/25 or 6/7.5).
* Mesopic pupil size measured with the Zywave II WaveFront Aberrometer must be < 7.0 mm and photopic pupil size measured with the Orbscan II/ IIz must be > 2.9 mm.

Additional Inclusion Criteria for Proscan Treatments

* For Proscan myopic subjects require a sphere between -0.5 D up to -10.0 D and cylinder between -0.5 D up to -4.0 D (not corneal astigmatism) and SE up to -12.0 D
* For Proscan hyperopic subjects require a sphere between +0.5 D up to +4.0 D and cylinder between +0.5 D up to +4.0 D (not corneal astigmatism) and SE up to +6.0 D.

Additional Inclusion Criteria for Zyoptix Treatments

For Zyoptix myopic subjects require a sphere between -0.5 D up to -10.0 D and cylinder between -0.5 D up to -4.0 D (not corneal astigmatism) and SE up to -12.0 D

* For Zyoptix hyperopic subjects require a sphere between +0.5 D up to +4.0 D and cylinder between +0.5 D up to +4.0 D (not corneal astigmatism) and SE up to +6.0 D.
* For all treatments with the Zyoptix algorithm, the high-order-aberration must be at least 0.35µm.

Additional Inclusion Criteria for Supracor Treatments

* For treatments with the SUPRACOR presbyopic algorithm, subjects have to be at least 45 years old and no more than 85 years
* Myopic subjects must have up to -7.0 diopters (D) of absolute spherical myopia (not spherical equivalent), with up to -4.0 D of refractive astigmatism (NOT corneal astigmatism) by manifest subjective refraction. The spherical equivalent and must be no more than -9.0 D.
* Hyperopic subjects must have up to +4 diopters (D) of absolute spherical hyperopia (not spherical equivalent), with up to +2.5 D of refractive astigmatism (NOT corneal astigmatism) by manifest subjective refraction in both eyes. The spherical equivalent must be no more than +5.25 D.
* Subjects must have presbyopia as determined by an age-related need for optical aid(> +1.50 D) for reading with their best distance correction and been screened success-fully for acceptance of the SUPRACOR simulation.

Exclusion Criteria

* Subjects for whom the combination of their baseline corneal thickness and the planned operative parameters for the LASIK procedure would result in less than 250 microns of remaining posterior corneal thickness below the flap postoperatively.
* Hyperopic eyes for which the baseline manifest subjective refraction exhibits a difference of greater than ± 0.75 D in sphere power, or a difference of greater than ± 0.50 D in cylinder power, or a difference in cylinder axis of more than 15 degrees compared to the baseline cycloplegic subjective refraction. For manifest cylinder of less than ±0.75 D, the differ-ence in cylinder axis would not be taken into consideration.
* Subjects with anterior segment pathology, including dry eye syndrome and cataracts, which in the Investigator's opinion would interfere with best spectacle-corrected visual acuity or a successful treatment.
* Subjects with evidence of retinal vascular disease. Subjects with any residual, recurrent, or active ocular disease, or corneal abnormality that in the Investigator's opinion would interfere with BSCVA or a successful treatment.
* Subjects with signs of keratoconus or Subjects with unstable central keratometry readings with irregular mires.
* Subjects who had previous intraocular or corneal surgery of any kind, including any type of Excimer laser surgery for either refractive or therapeutic purposes.
* Subjects who have a history of Herpes simplex or Herpes zoster keratitis or history of glaucoma or glaucoma suspect, corneal edema, or increased IOP > 22mmHg or risk for angle closure.
* Subjects immunocompromised or carrying diagnosis of connective tissue disease, clinically significant atopic disease, diabetes, autoimmune diseases and other acute or chronic illnesses that will increase the risk to the subject or confound the outcomes of this study.
* Subject taking systemic medications likely to affect wound healing such as corticosteroids or antimetabolites.
* Subjects who are known to be pregnant, lactating, or who plans to become pregnant over the course of the study.
* Subjects with an ocular muscle disorder including a strabismus or nystagmus, or other disorders affecting fixation.
* Subjects with cognitive impairments or other vulnerable persons.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
For Proscan and Zyoptix: - The percentage of treated eyes within +/- 0.50D of target refraction. For Supracor: - The percentage of treated eyes with a best corrected high contrast distance VA of Snellen 20/25 (6/7.5 or 0.1 logMAR) or better | Myopia: 6 months, Hyperopia 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ang, M.D., Principal Investigator — Asian Eye Institute
Locations (1):
- Asian Eye Institut, Manila, Philippines